CLINICAL TRIAL: NCT02636296
Title: The Effects of 12 Weeks Pilates-inspired Exercise Training on Functional Performance in Older Women: a Randomized Study
Brief Title: The Effects of 12 Weeks Pilates-inspired Exercise Training on Functional Performance in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ruth Caldeira de Melo, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HI017/2010
Record Dates: First submitted 2015-12-14; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Aging
Keywords: Pilates method; elderly; postural balance
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates (Experimental): Group received 12 week of inspired-Pilates intervention (2 days/week, 60 minutes duration).
  Interventions: Other: Pilates
- Control (Other): Control group was oriented to maintain the habitual activities during 12 weeks
  Interventions: Other: Control

INTERVENTIONS:
Other: Pilates — The Pilates program was conducted twice weekly, 60 minutes/session, for twelve consecutive weeks by a certified Pilates Instructor.
  Arms: Pilates
Other: Control — The control group did not receive the Pilates training program and were instructed to maintain their currently activities during the twelve-week follow-up period.
  Arms: Control

SUMMARY:
The purpose of the present study was to investigate the effects of 12-week Pilates-inspired exercise on functional performance in community-dwelling older women.

DETAILED DESCRIPTION:
Pilates is an exercise system developed over 70 years ago that has been recently received attention due to its beneficial effects on postural stability, coordination, muscle strength and flexibility. The studies published involving Pilates were very different among them regarding intervention period (5, 8, 12 and 24 weeks), frequency (2 and 3 sessions/week) and exercises (mat, mat with accessories, apparatus and others combinations), making meaningful comparison difficult. Furthermore, other important physical features to maintain an independent life at older age, such as cardiorespiratory fitness, were accessed in few studies. So, the effective benefits of Pilates method on physical fitness of community-dwelling older people remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* good health based on clinical examination (doctor's certificate)
* good functional capacity(physical examination)

Exclusion Criteria:

* current smokers
* obese (BMI >30 Kg/cm2)
* musculoskeletal limitations
* neurologic diseases
* cardiovascular diseases
* condition that contraindicated exercise
* regularly engaged in other physical conditioning program (>2x/week and/or >150min/week)

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
physical fitness | changes from baseline physical fitness at 12 weeks
  In this study, physical fitness includes strength, balance and aerobic resistance.